CLINICAL TRIAL: NCT03699748
Title: Lay Health Worker Engage, Educate, and Encourage Patients to Share
Acronym: LEAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 40447; K23MD013474-01 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: End of Life; Cancer
Keywords: cancer; end of life; patient-centered
MeSH Terms: conditions — Death; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Arm (Experimental): Patients randomized into the intervention will be assigned a lay health worker who will contact the patient to begin the intervention. The intervention includes: education on early advance care planning, documenting goals of care, assessing symptoms, and coordinating community services (such as home health, home visits, and home hospice).
  The intervention arm will also receive usual care as provided by Unite Here Health and their local oncologists.
  Interventions: Behavioral: Lay Health Worker Intervention; Other: Usual Care
- Control Group Arm (Active Comparator): The control group arm will receive usual care as provided by Unite Here Health and their local oncologists.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Lay Health Worker Intervention — Patients randomized into the intervention will be assigned a lay health worker who will contact the patient to begin the intervention. The intervention includes: education on early advance care planning, documenting goals of care, assessing symptoms, and coordinating community services (such as home health, home visits, and home hospice). The intervention is provided along with usual care as provided by Unite Here Health and local oncologists.
  Arms: Intervention Group Arm
Other: Usual Care — Usual care as provided by Unite Here Health and local oncologists

SUMMARY:
The purpose of the LEAPS program is to understand how a trained lay health worker who engages with newly diagnosed patients after a diagnosis of an advanced stage of cancer can help to engage patients in advance care planning, improve patient satisfaction with their decision-making, activation, quality of life, and healthcare resource utilization.

DETAILED DESCRIPTION:
Unite Here Health proposes to implement and evaluate several critical elements to be in alignment with the mission of the organization to provide high value care to their members. The Lay Health Worker Engages, Educates, and Encourages Patients to Share intervention is an innovative program that will strengthen provider-patient relationship and facilitate whole person care about matters important to Unite Here Health members who are diagnosed with cancer and important to support network and family. The project is intended to help establish Goals of Care Plan with appropriate documentation, develop, deploy, and evaluate a model of care for persons with cancer that is intended to improve clinical outcomes and experience of care for individuals. The intervention provides patients with lay health coaches who assist patients and their families in discussing goals of care and engage in shared-decision making. The goal of the project is to demonstrate that there is improved documentation of goals of care, patient experiences, patient activation and quality of life outcomes, and that the program helps to reduce utilization of health care resources at the end of life.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with a cancer diagnosis.
2. Patients with any relapse or progressive disease (any cancer diagnosis) as identified by imaging or biopsy and confirmed by physician.
3. The patients must be 18 years or older.
4. Patients must have the capacity to verbally consent.

Exclusion Criteria:

1. Inability to consent to the study due to lack of capacity as documented by the referring physician.
2. Patients without a newly diagnosed malignancy or patients without relapse of disease.
3. Patients not eligible for Fund benefits.

Patients without a newly diagnosed malignancy or patients without relapse of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manali I Patel, MD MPH MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel MI, Kapphahn K, Wood E, Coker T, Salava D, Riley A, Krajcinovic I. Effect of a Community Health Worker-Led Intervention Among Low-Income and Minoritized Patients With Cancer: A Randomized Clinical Trial. J Clin Oncol. 2024 Feb 10;42(5):518-528. doi: 10.1200/JCO.23.00309. Epub 2023 Aug 25. PMID 37625110
- [Derived] Patel MI, Khateeb S, Coker T. A randomized trial of a multi-level intervention to improve advance care planning and symptom management among low-income and minority employees diagnosed with cancer in outpatient community settings. Contemp Clin Trials. 2020 Apr;91:105971. doi: 10.1016/j.cct.2020.105971. Epub 2020 Mar 4. PMID 32145441

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Control Group: The control group arm participants receive usual care as provided by Unite Here Health and their local oncologists.
- Lay Health Worker Intervention Group: Patients randomized into the intervention are assigned a lay health worker who will contact the patient to begin the intervention, including: education on early advance care planning, documenting goals of care, assessing symptoms, and coordinating community services (such as home health, home visits, and home hospice). The intervention arm participants also receive usual care as provided by Unite Here Health and their local oncologists.
Period: Overall Study
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Started | 80 | 80
Completed Baseline Survey | 80 | 80
Completed 4 Month Survey | 74 | 71
Completed 12 Month Survey | 59 | 57
Completed | 58 | 57
Not Completed | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Control Group: The control group arm participants receive usual care.
- Lay Health Worker Intervention Group: Patients randomized into the intervention are assigned a lay health worker who will contact the patient to begin the intervention, and also receive usual care.
- Total: Total of all reporting groups
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 89] | 58 [21 to 80] | 58 [21 to 89]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 37 | 38 | 75
  Female | 42 | 41 | 83
  Non-binary | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 47
  Not Hispanic or Latino | 59 | 54 | 113
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 18 | 13 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 23 | 21 | 44
  White | 38 | 44 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 80 | 160
Annual household income [Count of Participants; unit: Participants]
  < $25,000 | 10 | 14 | 24
  ≥ $25,000 to $34,999.00 | 50 | 53 | 103
  ≥ $35,000 to $49,999.00 | 20 | 13 | 33
City [Count of Participants; unit: Participants] — Location where participant received care
  Participants
    Atlantic City, NJ | 53 | 55 | 108
    Chicago, IL | 27 | 25 | 52
Education Level [Count of Participants; unit: Participants]
  Less than high school | 61 | 68 | 129
  High school | 15 | 10 | 25
  2-year college or Bachelor degree | 4 | 2 | 6
Anatomic site of cancer diagnosis [Count of Participants; unit: Participants]
  Breast | 22 | 15 | 37
  Gastrointestinal | 16 | 14 | 30
  Genitourinary | 10 | 9 | 19
  Lung | 10 | 11 | 21
  Ovarian | 5 | 8 | 13
  Malignant hematologic | 7 | 11 | 18
  Head and Neck | 2 | 5 | 7
  Other (skin, soft tissue, brain) | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life Using the Functional Assessment of Cancer Therapy - General Survey
Description: Each patient will receive a quality of life survey (Functional Assessment of Cancer Therapy - General Survey) at baseline and 4 months. We will measure the change in quality of life at baseline to 4 months. Scores for quality of life will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G), a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Each question is a 5-point likert scale item. Scores range from 0-108. The higher the score, the better the quality of life.
Time Frame: Change in Quality of Life from Baseline to 4 Months
Population: Participants who completed the survey at each respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
score on a scale
  Baseline | 74.1 (16.5) | 73.5 (15.8)
  Month 4: number analyzed (Participants) | 74 | 71
  Month 4 | 70.3 (16.8) | 80.7 (16.4)
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; p < 0.001, Type III F test; Mean Difference (Net) = 10.92, 95% CI 2-sided [7.27 to 14.58]

2. Secondary Outcome: Patient Satisfaction With Decision-Making Using the Satisfaction With Decision (SWD) Survey
Description: The validated Satisfaction with Decision (SWD) Survey was administered to all participants at 4 months after study enrollment. The SWD is a 6-item questionnaire, where respondents rate their agreement with 6 statements (e.g. "I am satisfied that I am adequately informed about the issues important to my decision") on a likert-type scale. Answer options were (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree. Responses to each item were averaged to give a score of 0 to 5 where 0 indicated lowest satisfaction and 5 indicated most satisfied with decision making. Scores for each group were averaged at 4 months after study enrollment. Results are expressed as a proportion of participants who responded "strongly agree" at 4 months post-enrollment on the SWD scale, which measured ratings of decision-making. Changes in the proportion of participants who responded "strongly agree" are reflected from baseline to 4 months post-enrollment.
Time Frame: Proportion of patients who strongly agree that decisions about their health care were theirs to make at 4 months post study enrollment.
Population: At 4 Months, 74 (92.5%) in the control group and 71 (88.8%) in the intervention group completed this survey and 6 (7.5%) participants in the control group and 9 (11.3%) participants in the intervention group had died by the time of this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 74 | 71
Participants | 23 | 64

3. Secondary Outcome: Patient Satisfaction With Decision-Making Using the Satisfaction With Decision Survey
Description: The validated Satisfaction with Decision (SWD) Survey was administered to all participants at 12 months after study enrollment. The SWD is a 6-item questionnaire, where respondents rate their agreement with 6 statements (e.g. "I am satisfied that I am adequately informed about the issues important to my decision") on a likert-type scale. Answer options were (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree. Responses to each item were averaged to give a score of 0 to 5 where 0 indicated lowest satisfaction and 5 indicated most satisfied with decision making. Scores for each group are averaged at 12 months after study enrollment. Results are expressed as a proportion of participants who responded "strongly agree" at 12 months post-enrollment on the SWD scale, which measured ratings of decision-making. Changes in the proportion of participants who responded "strongly agree" are reflected from baseline to 12 months.
Time Frame: Proportion of patients who strongly agree that decisions about their health care were theirs to make at 12 months post study enrollment.
Population: A total of 59 participants (73.8%) in the control group and 56 (70.0%) in the intervention group completed this survey question at 12-months post study enrollment; 21 (26.3%) participants in the control group and 23 (28.8%) participants in the intervention group had died at the time of the 12-month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 59 | 56
Participants | 16 | 48

4. Secondary Outcome: Patient Activation Using the Patient Activation Measure Survey
Description: Each patient will receive the 13-item Patient Activation Measure (PAM-13) at 4 months after study enrollment. This is a validated measure from Insignia Health. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-13, minimum score is 0 and maximum is 100. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining Behaviors and Pushing Further. Scores for each group will be averaged at 4 months after study enrollment.
Time Frame: Change in Patient Activation Measure from baseline to 4 months post enrollment.
Population: Missingness was only observed due to death among 6 (7.5%) participants in the control group and 9 (11.3%) participants in the intervention group who had died prior to the 4-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 74 | 71
score on a scale
  Baseline | 53.5 (10.3) | 53.4 (9.80)
  4 Months | 53.3 (10.1) | 65.9 (14.7)
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate for 4 Months = 12.88 — 12.88 (9.49 - 16.28); Effect estimates were expected mean differences in Patient Activation Measure scores between groups from baseline. Effect estimates were estimated using generalized estimating equations (GEE) models as a function of treatment group, categorical time (baseline, 4 months and 12 months), and an interaction term between treatment group and time with an exchangeable correlation clustered within person. The effect estimate column shows the difference between change in the intervention group from baseline and the change in the control group from baseline

5. Secondary Outcome: Patient Activation Using the Patient Activation Measure Survey
Description: Each patient will receive the 13-item Patient Activation Measure (PAM-13) at 12 months after study enrollment. This is a validated measure from Insignia Health. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-13, minimum score is 0 and maximum is 100 (highest level of activation). Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining Behaviors and Pushing Further. Scores for each group will be averaged 12 months after study enrollment.
Time Frame: Change in Patient Activation Measure from baseline to 12 months post-enrollment.
Population: Missingness was only observed due to death among 21 (26.3%) participants in the control group and 23 (28.8%) participants in the intervention group who had died prior to this 12-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 58 | 57
score on a scale | 57.6 (10.8) | 77.7 (11.2)
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate for 12 Months = 20.65 — 20.65 (6.97 - 24.32); Effect estimates were expected mean differences in Patient Activation Measure scores between groups from baseline. Effect estimates were estimated using generalized estimating equations (GEE) models as a function of treatment group, categorical time (baseline, 4 months and 12 months), and an interaction term between treatment group and time with an exchangeable correlation clustered within person

6. Secondary Outcome: Patient Quality of Life Using the Functional Assessment of Cancer Therapy - General Survey
Description: Each patient will receive a quality of life survey (Functional Assessment of Cancer Therapy - General Survey) at 12 months. Scores for quality of life will be assessed using the Functional Assessment of Cancer Therapy - General Survey-General survey. The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Each question is a 5-point likert scale item. Scores range from 0-108. The higher the score, the better the quality of life.
Time Frame: Health-related quality of life at 12 months
Population: Participants who completed the survey at 12 months are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 59 | 57
score on a scale | 73.3 (15.6) | 84.4 (16.5)
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; p = 0.001, Type III F-test; Median Difference (Net) = 11.05, 95% CI 2-sided [7.09 to 15.00]

7. Secondary Outcome: Emergency Department Visit (Chart Review)
Description: Emergency Department Use for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Population: All enrolled participants
Measure: Number; unit: Emergency Department Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Emergency Department Visits | 15 | 12

8. Secondary Outcome: Emergency Department Visit (Chart Review)
Description: Emergency Department Use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Number; unit: Emergency Department Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Emergency Department Visits | 24 | 27
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 0.91 — 0.91 (0.40-2.09); Odds Ratios for any emergency room use and any hospitalization use were estimated using logistic regression models

9. Secondary Outcome: Emergency Department Visit (Chart Review)
Description: Emergency Department Use will be abstracted by electronic medical record chart review for each patient who is deceased within 12 months of enrollment, looking at their ER visits during the last 30 days of life.
Time Frame: Last 30 days of life up to 12 months from patient enrollment
Population: Sample of 21 participants in the control group and 23 participants in the intervention group who died within 12 months of study enrollment.
Measure: Number; unit: Emergency Department Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 21 | 23
Emergency Department Visits | 3 | 1
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 0.27 — 0.27 (0.03 - 2.85); Odds Ratios for any ED Use were estimated using logistic regression models

10. Secondary Outcome: Hospitalization Visit (Chart Review)
Description: Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Number; unit: Hospital Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Hospital Visits | 16 | 32
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 0.38 — 0.38 (0.18-0.76); Odds Ratios for any emergency room use and any hospitalization use were estimated using logistic regression models

11. Secondary Outcome: Hospitalization Visits (Chart Review)
Description: Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after study enrollment
Measure: Number; unit: Hospital Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Hospital Visits | 50 | 33
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 0.42 — 0.42 (0.22-0.79); Odds Ratios for any emergency room use and any hospitalization use were estimated using logistic regression models

12. Secondary Outcome: Hospitalization Visits (Chart Review)
Description: Hospitalization use will be abstracted by electronic medical record chart review for each patient who is deceased within12 months of enrollment, looking at their hospital visits during the last 30 days of life.
Time Frame: last 30 days of life
Population: as for outcome 9
Measure: Number; unit: Hospital Visits
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 21 | 23
Hospital Visits | 3 | 6
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 0.38 — 0.38 (0.08-1.75); Odds Ratios for Hospitalization Use were estimated using logistic regression models

13. Secondary Outcome: Advance Directive Documentation (Chart Review)
Description: Advance Directive documentation for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants
  Baseline | 1 | 0
  4 Months | 15 | 46
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio, log = 5.86 — Odds Ratios for Goals of Care Documentation, Advance Directive Documentation, and Physician Order for Life Sustaining Treatment Documentation were estimated based on assessments 4-months and 12-months post-enrollment with logistic regression

14. Secondary Outcome: Advance Directive Documentation (Chart Review)
Description: Advance Directive documentation for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 55 | 72
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 4.09 — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Physician Orders for Life Sustaining Treatment (Chart Review)
Description: Physician Orders for Life Sustaining Treatment (POLST) documentation for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 5 | 25
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 6.82 — 6.82 (2.46-18.93); Odds Ratios for Physician Order for Life Sustaining Treatment Documentation were estimated based on assessments 4-months post-enrollment with logistic regression

16. Secondary Outcome: Physician Orders for Life Sustaining Treatment (Chart Review)
Description: Physician Orders for Life Sustaining Treatment (POLST) documentation for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 13 | 33
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 3.62 — 3.62 (1.73-7.60); Odds Ratios for Physician Order for Life Sustaining Treatment Documentation were estimated based on assessments at 12-months post-enrollment with logistic regression

17. Secondary Outcome: Goals of Care Documentation (Chart Review)
Description: Goals of Care documentation for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 10 | 44
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio, log = 8.56 — [estimate comment as in outcome 13, analysis 1]

18. Secondary Outcome: Goals of Care Documentation (Chart Review)
Description: Goals of Care documentation for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 23 | 71
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio, log = 19.55 — Odds Ratios for Goals of Care Documentation, Advance Directive Documentation, and Physician Order for Life Sustaining Treatment Documentation were estimated based on assessments at 12-months post-enrollment with logistic regression

19. Secondary Outcome: Total Costs of Care
Description: Total Costs of Care will be evaluated by review of claims data from time of enrollment until 12 months post-enrollment
Time Frame: 12 months after patient enrollment
Measure: Median (Inter-Quartile Range); unit: US Dollars
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
US Dollars | 153,980.60 [52,612.08 to 243,751.00] | 72,585.06 [23,601.07 to 150,670.06]
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate = 0.65 — 0.65 (0.44-0.98); Proportional change in total health care costs are expressed as referent to the control group and were modeled using a generalized linear model with gamma link-log function to account for skewed cost data after adjustment for length of follow-up

20. Secondary Outcome: Total Costs of Care End of Life
Description: Total Costs of Care during the last 30 days of life will be evaluated by review of claims data from the 30 days preceding death for those patients who become deceased within 12 months of study enrollment.
Time Frame: Last 30 days of life up to 12 months from patient enrollment
Population: as for outcome 9
Measure: Number; unit: US Dollars
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 21 | 23
US Dollars | 6,211 | 5,471
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate = 0.57 — 0.57 (0.28 - 1.18); Proportional change in total health care costs are expressed as referent to the control group and were modeled using a generalized linear model with gamma link-log function to account for skewed cost data

21. Secondary Outcome: Palliative Care Use (Chart Review)
Description: Palliative Care Use for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 5 | 25
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 6.82 — 6.82 (2.46-18.93); Odds Ratios for palliative care receipt and hospice receipt were estimated based on assessments 4-months and 12-months post-enrollment compared with baseline (time of enrollment) using logistic regression

22. Secondary Outcome: Palliative Care Use (Chart Review)
Description: Palliative Care Use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 13 | 33
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 3.62 — 3.62 (1.73-7.60); [other analysis details as in outcome 21, analysis 1]

23. Secondary Outcome: Palliative Care Use (Chart Review)
Description: Palliative Care Use will be abstracted by electronic medical record chart review for each patient who is deceased within12 months of enrollment, looking at their palliative care usage during the last 30 days of life.
Time Frame: last 30 days of life
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 21 | 23
Participants | 6 | 16
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate = 5.71 — 5.71 (1.56-20.93); Odds Ratios for any ED Use and any Palliative Care were estimated using logistic regression models. Incidence Rate Ratios (IRR) were estimated using Poisson models. All ratios are expressed as referent to the control group

24. Secondary Outcome: Hospice Use (Chart Review)
Description: Hospice Use for each patient will be abstracted by electronic medical record chart review for each patient at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 2 | 8
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 4.33 — 4.33 (0.89-21.08); [other analysis details as in outcome 21, analysis 1]

25. Secondary Outcome: Hospice Use (Chart Review)
Description: Hospice Use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 80 | 80
Participants | 6 | 16
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Odds Ratio (OR) = 2.76 — 2.76 (1.01-7.55); Odds Ratios for palliative care receipt and hospice receipt were estimated based on assessments at 12-months post-enrollment compared with baseline (time of enrollment) using logistic regression

26. Secondary Outcome: Hospice Use (Chart Review)
Description: Hospice Use will be abstracted by electronic medical record chart review for each patient who is deceased within12 months of enrollment, looking at their hospice use during the last 30 days of life.
Time Frame: last 30 days of life
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 21 | 23
Participants | 6 | 16
Statistical Analysis 1: Comparison: Usual Care Control Group vs Lay Health Worker Intervention Group; Test type: Other; Effect Estimate = 5.71 — 5.71 (1.56-20.93); Odds Ratios for any ED Use and any Hospice Receipt were estimated using logistic regression models. Incidence Rate Ratios (IRR) were estimated using Poisson models. All ratios are expressed as referent to the control group

27. Secondary Outcome: Survival (Chart Review)
Description: Survival rate for patients will be abstracted by electronic medical record chart review at 4 months after enrollment.
Time Frame: 4 months after patient enrollment
Reporting Status: Not Posted

28. Secondary Outcome: Survival (Chart Review)
Description: Survival rate for patients will be abstracted by electronic medical record chart review at 12 months after enrollment.
Time Frame: 12 months after patient enrollment
Reporting Status: Not Posted

29. Secondary Outcome: Patient Satisfaction With Decision-Making Using the Satisfaction With Decision Survey
Description: The validated Satisfaction with Decision (SWD) Survey was administered to all participants at baseline. The SWD is a 6-item questionnaire, where respondents rate their agreement with 6 statements (e.g. "I am satisfied that I am adequately informed about the issues important to my decision") on a likert-type scale. Answer options were (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree. Responses to each item were averaged to give a score of 0 to 5 where 0 indicated lowest satisfaction and 5 indicated most satisfied with decision making. Results are expressed as a proportion of participants who responded "strongly agree" at Baseline on the Satisfaction with Decision scale, which measured ratings of decision-making.
Time Frame: Proportion of patients who strongly agreed the decisions about their health care were theirs to make at baseline (study enrollment).
Population: 79 (98.8%) participants in the control group and 80 (100%) participants in the intervention group completed this survey at time of enrollment in the study (baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
Number analyzed (Participants) | 79 | 80
Participants | 41 | 38

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Care Control Group | Lay Health Worker Intervention Group
All-Cause Mortality (participants affected / at risk) | 21/80 | 23/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03699748/Prot_SAP_000.pdf